CLINICAL TRIAL: NCT02667145
Title: Self-care Program Evaluation With Focus on Assistive Devices for Individuals With Hand Osteoarthritis
Brief Title: Assistive Device for Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Salgado Amaral (Other)
Responsible Party: Sponsor-Investigator, Daniela Salgado Amaral, Terapeuta Ocupacional, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFPernambuco2015
Record Dates: First submitted 2015-04-15; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hand Osteoarthritis
Keywords: hand osteoarthritis; self care program; assistive tecnology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Self care program focusing on the assistive device, For 4 weeks (1 to week lasting 90 minutes).
  Interventions: Other: Self care program focusing on the assistive device
- Control group (No Intervention): receive only a brochure with orientations of joint protection.

INTERVENTIONS:
Other: Self care program focusing on the assistive device — self-heed program focusing on the assistive device will consist of four weekly meetings lasting approximately 90 minutes. it will be stimulated the self-heed through knowledge of pathology and guidelines of protection articulate, and will be supplied, and trained the use of assistive devices to improve the performance of volunteers in their daily activities. Assistive devices are devices, not attached to the body, which help people with limited movements and restrictions on participation in the activities of everyday life. Example: thickening of tableware, tin openers. These volunteers will be evaluated in three stages: 1-initial assessment 2-after completion of the program and 90 days after the initial assessment. The questionnaires that will be used are: EVA; SACRAH; COPM; WHOQOL-Bref.
  Arms: Intervention

SUMMARY:
Randomized clinical trial , blind for evaluators, to assess the effectiveness of a self-care program using assistive technology for treatment of hand osteoarthritis.

DETAILED DESCRIPTION:
This program aims to:

* Encourage the use of assistive devices on a daily basis as the main form of joint protection.
* Encourage individual motivation, from the group in attendance, behavior change, developing the capacity of self-management of individuals of their health problems.

Will be held for 4 meetings with an average duration of 90 minutes. Meeting 1: Its proposal address the importance of self-care in the treatment of chronic diseases; knowing the OA of the hands and their main characteristics; recognize the importance of hand function for carrying out activities; understand the meaning of self-care and joint protection; motivation adherence to the program and behavior change.

Meeting 2: Present assistive devices as a protection feature; teach joint protection techniques and energy conservation focusing on the assistive device; deliver and demonstrate the use of assistive devices.

Meeting 3:Encouraging the adhesion of the techniques presented; making workshop for daily activities; verify the difficulties with devices use by the volunteers.

Meeting 4: Strengthening guidance given in previous meetings; make closing with the group to in connection with the program; motivated to continue carrying out the activities at home.

ELIGIBILITY:
Inclusion Criteria:

* Hand OA diagnosis according to the criteria of the American College of Rheumatology (ACR )
* Be properly registered in the rheumatology clinic of Hospital das Clínicas

Exclusion Criteria:

* Surgical treatment or infiltration in the hands, in the last 6 months;
* Treatment of occupational therapy and / or physical therapy, or use of any TA feature (assist device or stent) in the last 6 months;
* Diagnosis of another rheumatologic disease or musculoskeletal system that compromise the hands associated.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Occupational Performance | 4 weeks
  involvement of daily activities by the Canadian Occupational Performance Measure (COPM)

SECONDARY OUTCOMES:
Quality of life | 4 weeks
  Evaluation by WHO-QOL bref
Manual functional | 4 weeks
  Evoluation by SACRAH
Pain | 4 weeks
  Evaluation by visual analogue pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Claudia DL Marques, PhD, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Hospital das Clínicas - Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Derived] Amaral DS, Duarte ALBP, Barros SS, Cavalcanti SV, Ranzolin A, Leite VMM, Dantas AT, Oliveira ASCRC, Santos PS, Silva JCA, Marques CDL. Assistive devices: an effective strategy in non-pharmacological treatment for hand osteoarthritis-randomized clinical trial. Rheumatol Int. 2018 Mar;38(3):343-351. doi: 10.1007/s00296-017-3892-1. Epub 2017 Nov 28. PMID 29185087